CLINICAL TRIAL: NCT04570085
Title: Multicentre, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Effect of a 30-week Caffeine Treatment on Cognition in Alzheimer's Disease at Beginning to Moderate Stages
Brief Title: Effect of CAFfeine on Cognition in Alzheimer's Disease
Acronym: CAFCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other); Laboratory of excellence DISTALZ (Unknown); Région Nord-Pas de Calais, France (Other); Meo coffee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018_95; 2019-002360-27 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-09-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; caffeine; cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): after a 3 weeks up titration period, 1 capsule of 200 mg twice a day during 27 weeks (ie 400mg/day)
  Interventions: Drug: Caffeine
- placebo (Placebo Comparator): after a 3 weeks up titration period, 2 capsules per day during 27 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — 100mg caffeine capsule treatment, beginning after caffeine diet during 6 weeks, titrate in 3 weeks (by 100mg stages) until 400mg aim dose per day in 2 doses during 27 weeks, and finally interrupt according to the same negative titration.
  Arms: Caffeine
Drug: Placebo — Placebo capsule treatment, beginning after caffeine diet during 6 weeks, titrate in 3 weeks until 2 doses aim dose per day during 27 weeks, and finally interrupt according to the same negative titration.
  Arms: placebo

SUMMARY:
Sporadic Alzheimer's disease is a multifactorial illness arising a major medico-economic stakes for our aging societies. There is currently no curative treatment available.

Coffee is a complex beverage with psychostimulant properties whose main effective element, caffeine, has a pleiotropic effect on the central nervous system. Caffeine pharmacological properties enable its use like an Alzheimer's disease symptomatic treatment. Its supposed benefits mustn't obscure anxiety and insomnia caffeine effect at large dose, which Alzheimer's patients might be more vulnerable.

The main study objective is to evaluate placebo-controlled caffeine efficacy (30 treatments weeks) on cognitive decline in Alzheimer's disease dementia at beginning to moderate stage (MMSE 16-24).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 at screening
* Probable Alzheimer dementia according to the criteria of the National Institute on Aging-Alzheimer's Association; diagnosis must be supported by brain imaging (CT or MRI) and blood test (including ionogram, kidney and liver function, calcemia, CRP, TSH, B12 vitamins and folates) performed in routine care
* MMSE score ≥16
* Presence of an informant and caregiver, living with the patient
* IAChE and/or Memantine treatment non-compulsory ; If implemented it must be effective and stable for 2 months before the selection visit and must remain stable for the duration of the study

Exclusion Criteria:

* Patients who refuse to adopt a low caffeine diet (eviction of tea, caffeinated sodas, chocolate in large quantities)
* Current major depressive episode according to DSM-5 criteria
* Another chronic pathology of the central nervous system
* Major anxiety according to the clinician (consistent with the corresponding nPI-R items that must indicate a severity >2 and an impact >3)
* Sleep disorders defined by severity and an impact on NPI-R; a patient fitted for OSA may be included if the device has been in use for 3 months and well tolerated (stable)
* Decompensated heart disease or severe rhythm disorder (excluding slow, treated and stable chronic atrial fibrillation)
* Active smoking
* For childbearing women : pregnancy in progress or planned (A pregnancy test will be performed)
* Patients who take forbidden treatment :

  * Psychotropic treatments introduced or modified < 2 months before inclusion
  * Chronic use of CYP1A2 inducing or inhibiting drugs
  * All caffeine-containing specialties
  * Drugs that influence caffeine metabolism
  * Drugs that may interact with caffeine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes in NTB scores | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment

SECONDARY OUTCOMES:
Caffeine treatment effect on MMSE score | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on MMSE score
Caffeine treatment effect on NTB subscores | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on NTB subscores
Caffeine treatment effect on TAP scores | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on TAP scores
Caffeine treatment effect on Epworth score | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on Epworth score
Caffeine treatment effect on DAD-6 score | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on DAD-6 score
Caffeine treatment effect on QoL-AD score | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on QoL-AD score
Caffeine treatment effect on CGIC score | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on CGIC score
Caffeine treatment effect on Zarit score | 30 weeks after randomization
  difference between randomized value and value after 30 weeks of treatment on Zarit score
persistent effect of caffeine treatment on MMSE score after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on MMSE score
persistent effect of caffeine treatment on NTB subscores after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on NTB subscores
persistent effect of caffeine treatment on TAP scores after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on TAP scores
persistent effect of caffeine treatment on Epworth score after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on Epworth score
persistent effect of caffeine treatment on DAD-6 score after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on DAD-6 score
persistent effect of caffeine treatment on QoL-AD score after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on QoL-AD score
persistent effect of caffeine treatment on Zarit score after a 6 weeks wash out period | 36 weeks after randomization
  difference between value after 30 weeks of treatment and value after a 6 weeks wash out period (from Week 30 to Week 36) on Zarit score
Caffeine effect heterogeneity: impact of AD treatment | 30 weeks after randomization
  impact of AD treatment on caffeine effect
Caffeine effect heterogeneity: impact of ApoE4 status | 30 weeks after randomization
  impact of ApoE4 status on caffeine effect
Caffeine effect heterogeneity: impact of caffeine metabolism speed | 30 weeks after randomization
  impact of caffeine metabolism on caffeine effect
Caffeine effect heterogeneity: impact of gender | 30 weeks after randomization
  impact of gender on caffeine effect
Caffeine safety profile: NPI scores | 30 weeks after randomization
  changes in NPI scores and subscores between caffeine and placebo arms
Caffeine safety profile: heart beat | 30 weeks after randomization
  changes in heart beat between caffeine and placebo arms
Caffeine safety profile: blood pressure | 30 weeks after randomization
  changes in blood pressure between caffeine and placebo arms
Caffeine and its derivatives concentrations in blood samples | 30 weeks after randomization
  increase in caffeinemia and its derivatives in the morning (fasting samples)

CONTACTS AND LOCATIONS:
Overall Officials: thibaud LEBOUVIER, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (17):
- France (17):
  - CHU Amiens, Amiens
  - CH Arras, Arras
  - CH Beauvais, Beauvais
  - CH Béthune, Béthune
  - CHU Caen, Caen
  - CH Calais, Calais
  - CH Dunkerque, Dunkirk
  - CH Le Quesnoy, Le Quesnoy
  - CH Lens, Lens
  - Hôpital Roger Salengro, Lille
  - CHU Lille consultation mémoire Les Bâteliers, Lille
  - CH Roubaix, Roubaix
  - CHU Rouen, Rouen
  - CH Saint Quentin, Saint-Quentin
  - CH Seclin, Seclin
  - CH Tourcoing, Tourcoing
  - CH Valenciennes, Valenciennes